CLINICAL TRIAL: NCT04514263
Title: Evaluation of the Post-surgical Discomfort in Patients Undergoing Diagnostic Oral Biopsies
Brief Title: Oral Biopsies: Evaluation of the Post-surgical Discomfort
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Carlo Lajolo, Associate Professor, Catholic University of the Sacred Heart
Other Study IDs: OHIP-OB
Record Dates: First submitted 2020-08-06; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Quality of Life; Biopsy Wound; Surgical Wound; Healing Surgical Wounds
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oral Biopsy: Patients with oral lesions undergoing diagnostic or therapeutic biopsies either for benign lesions or potentially malignant disorders or malignant lesions or salivary glands diseases.
  Interventions: Other: OHIP-14 Administration; Other: VNS Administration

INTERVENTIONS:
Other: OHIP-14 Administration — All patients fulfilled the OHIP-14 questionnaire three times: six hours, seven days and twenty-one days after the biopsy
Other: VNS Administration — All patients fulfilled the VNS scale three times: six hours, seven days and twenty-one days after the biopsy

SUMMARY:
Aim of this study is to evaluate the post-operative course in patients undergoing diagnostic or therapeutic oral mucosal biopsies.

To evaluate the wound healing, all variables connected with the surgery (including post-operative complications) were recorded. To evaluate the psychological and behavioral impact of the post-operative discomfort, two survey tools were administered: OHIP-14 and visual number scale of pain (VNS) were administered at 6h, 7 days and 21 days after biopsy.

ELIGIBILITY:
Inclusion Criteria:

* no systemic or local contraindications for surgical treatment
* need for an oral biopsy (both excisional and incisional).

Exclusion Criteria:

Since no absolute contraindications to oral biopsies are reported, no exclusion criteria were selected for this study, but if any relative contraindication was present (i.e. bleeding disorders) biopsy was performed after the resolution of the problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eighty-four patients were enrolled in this study; four of them were excluded because the clinical records were incomplete. Among the 80 patients left, 30 were males and 50 females, with a mean age of 60.25 years (range 23-88); clinical data about remote pathological history were collected: 31/80 patients did not have any systemic diseases, 22/80 only one disease, 27/80 more than one disease; 36/80 patients did not take any drug, 16/80 only one and 28/80 more than one; 63/80 patients did not smoke, 10/80 were former smokers and 7/80 were smokers.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-12-08 (Actual)

PRIMARY OUTCOMES:
Correlation between the clinical healing and patient perception | Six hours after an oral biopsy
  To evaluate whether the clinical evaluation of a wound healing shows a correspondence with the patient perception of the same process.
Correlation between the clinical healing and patient perception | One week after an oral biopsy
  To evaluate whether the clinical evaluation of a wound healing shows a correspondence with the patient perception of the same process.
Correlation between the clinical healing and patient perception | Three weeks after an oral biopsy
  To evaluate whether the clinical evaluation of a wound healing shows a correspondence with the patient perception of the same process.

SECONDARY OUTCOMES:
Correlation between OHIP-14 and VNS scale | Six hours after an oral biopsy
  Correlation between two different tools evaluating patient perception
Correlation between OHIP-14 and VNS scale | One week after an oral biopsy
  Correlation between two different tools evaluating patient perception
Correlation between OHIP-14 and VNS scale | Three weeks after an oral biopsy
  Correlation between two different tools evaluating patient perception
Clinical variables which influence the healing and patient perception | Six hours after an oral biopsy
  To evaluate which clinical variable (systemic or local) can modify the wound healing or the patient perception.
Clinical variables which influence the healing and patient perception | One week after an oral biopsy
  To evaluate which clinical variable (systemic or local) can modify the wound healing or the patient perception.
Clinical variables which influence the healing and patient perception | Three weeks after an oral biopsy
  To evaluate which clinical variable (systemic or local) can modify the wound healing or the patient perception.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of the Sacred Heart, Rome, Italy